CLINICAL TRIAL: NCT05949983
Title: Health Economic Evaluation of an Adapted Physical Activity Program for Women With Breast Cancer During the Active Phase of Treatment: a Randomized Controlled Trial
Brief Title: Health Economic Evaluation of an Adapted Physical Activity Program for Women With Breast Cancer
Acronym: EMEAPA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RC31/21/0339; 2022-A00017-36 (Other: ID-RCB)
Record Dates: First submitted 2023-06-13; First posted 2023-07-18 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Breast Neoplasm
Keywords: Physical Activity; Exercise; Exercise Therapy; Breast Neoplasms; Medical costs; Healthcare Costs
MeSH Terms: conditions — Breast Neoplasms; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- APA program Group (Experimental): patients treated and monitored for breast cancer under the APA programme
  Interventions: Other: APA Program
- Physical activity recommendation Group (Active Comparator): patients treated and monitored for breast cancer who have received recommendations for physical activity
  Interventions: Other: Recommendations for physical activity

INTERVENTIONS:
Other: APA Program — Patients treated and monitored for their breast cancer following the 6-month APA program.
  Arms: APA program Group
Other: Recommendations for physical activity — Patients treated and monitored for their breast cancer who have received recommendations for physical activity as well as a 6-month activity schedule. To facilitate patient acceptance and participation in this study, patients who will be randomized to the control group will be offered to follow the APA program after one year of inclusion
  Arms: Physical activity recommendation Group

SUMMARY:
Adapted physical activity (APA) was recognized as a non-drug therapy by the French Health Authority (HAS) in 2011. Very few studies have examined the efficiency of APA programs during the active phase of treatment in cancer patients. The investigators assumed that non-drug therapy such as APA could improve the quality of life and reduces health costs. The main objective of this study is to assess the efficiency of a standardized APA program, as compared to conventional management including simple recommendations for the practice of physical activity in women in phase active breast cancer treatment.

DETAILED DESCRIPTION:
Scientific rationale: The incidence of breast cancer in women is on the rise again over the period 2010-2018. The overall cost of cancer treatment is 16.8 billion euros, including 3.6 billion for drugs alone. The treatments are more and more prolonged, the proportion of anticancer drugs continues to increase with 10% of the amount reimbursed for drugs delivered in pharmacies in 2017.

Adapted physical activity (APA) was recognized as a non-drug therapy by the HAS in 2011. It reduces certain side effects of treatments, as well as certain symptoms linked to the catabolic activity of the disease such as: fat gain, loss of muscle mass, physical deconditioning, fatigue or pain. For breast cancer, a meta-analysis showed that APA following adjuvant therapy may have a beneficial effect on quality of life. The APA shows in particular for breast cancer, a reduction in all-cause mortality as well as specific mortality and a reduction in recurrence.The prescription of APA has been allowed since the 2016 health law but there is no coverage by the French national health insurance fund (CNAM) despite the benefits shown. APA is only accessible in a few centers in France that have chosen to offer it to patients, thus creating social inequalities in health.

Very few studies have examined the efficiency of APA programs during the active phase of treatment. They related to cohorts of 60 to 165 patients and uses different methods. The investigators decided to set up a study that can measure the efficiency of the standardized APA programs offered to patients diagnosed with breast cancer, assuming that non-drug therapy such as APA would improve the quality of life while reducing health costs.

Description of the procedures: The intervention consists of an initial consultation appointment with a medical check-up and physical tests, then inclusion in the standardized APA program for 6 months. The control group will be offered the same initial consultation appointment with medical check-up and physical tests and will receive recommendations for physical practice as well as a calendar of activities to be practiced independently for 6 months. Inclusion in the APA program will be offered one year after inclusion.

Follow-up: The data will be collected at T0, T + 3 months, T + 6 months, T + 9 months and T + 12 months in both arms. There will be 1 year of data analysis.

ELIGIBILITY:
Inclusion Criteria:

* women with breast cancer
* any type of breast cancer, all grades, all stages
* during treatment: surgery +/- chemotherapy +/- radiotherapy +/- hormone therapy

Exclusion Criteria:

* World Health Organization (WHO) 4
* Unstable angina
* Uncontrolled Atrial fibrillation
* Uncontrolled high blood pressure
* Recent myocardial infarction or myocarditis or pericarditis or thromboembolic disease (less than 3 weeks)
* Aortic stenosis or valve disease to operate
* Cardiac or respiratory failure, with dyspnea at rest
* Symptomatic anemia, thrombocytopenia
* Lytic or painful bone metastases, Severe osteoporosis
* Severe infectious syndrome,
* Surgery in the last 3 weeks
* Extreme fatigue, sharp pain, dizziness, disturbance of consciousness, severe undernutrition
* Contraindication to the practice of an adapted physical activity programme
* Currently involved or exclusion period of a interventional study or adapted Physical Activity program
* Patient with protective measures (guardianship, curators, and deprivation of liberty).
* Pregnancy or breastfeeding
* Patient with severe functional limitations

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 866 (Estimated)
Dates: Start 2024-12-23 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Comparison of physical activity programmes | 12 months
  Evaluation of the differential cost-utility ratio (cost / QALY), according to the perspective of the community over a 12-month period, of an adapted physical activity program (APA) in comparison to conventional care, including simple recommendations for physical activity for patients with breast cancer during the active phase of treatment.

SECONDARY OUTCOMES:
Breast cancer-specific quality of life | 12 months
  Breast Cancer Specific Quality of Life Questionnaire (QLQ) (BR23-QLQ-C30) is a 52-item questionnaire. The choices range from 1 "not at all" to 4 "very much".
Clinical efficacy | 12 months
  Progression-free survival measured for non-metastatic (relapse-free survival) and metastatic (progression-free survival) patients
Efficacy on specific functions | 12 months
  BR23-QLQ-C30 questionnaire.
  Breast Cancer Specific Quality of Life Questionnaire (BR23-QLQ-C30) is a 52-item questionnaire. The choices range from 1 "not at all" to 4 "very much".
Society impact (interview) | 12 months
  Zarit-Burden Interview
Society impact | 12 months
  Number of hours of informal help for basic and instrumental activities of daily life
Patient satisfaction | 12 months
  Patient satisfaction questionnaire (EORTC-IN-PATSAT32) is a 32-item questionnaire. The choices range from 1 "bad" to 4 "excellent".
Programme compliance rate | 12 months
  Traced by the reservation system for adapted physical activity (APA) sessions
Rate of hospital care | 12 months
  Direct medical costs
Rate of difference in the effect of the programme | 12 months
  Socioeconomic determinants (changes in income, socio-professional category, level of education and family environment)
Rate of financial benefit of the programme | 5 years
  Annual and 5-year net financial benefit of the systematic implementation of an adapted physical activity (APA) program

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Eve Rougé-Bugat, MD, Principal Investigator — University Toulouse
Locations (1):
- Marie-Eve Rougé-Bugat, Toulouse, France